CLINICAL TRIAL: NCT06281002
Title: Assessment of Accuracy of Full Digital Workflow in Fabrication of Four-Implant Screw-Retained Mandibular Hybrid Prostheses
Brief Title: Trueness of Full Arch Scans and Generated Digital Implant Models
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Omnia Hafez Mohamed, Clinical general dentist at MOH, Master degree candidate in oral and maxillofacial prosthodontics, Ain Shams University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-RecIM112323
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Denture; Complete Edentulism
Keywords: Intraoral scanning; Digital implant models; Edentulous mandible; Screw retained prosthesis; Geometric scanning aids

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional physical impressions (Active Comparator): Nine physical open tray impressions will be poured into a hard dental stone to obtain nine definitive implant casts with conventional implant analogs.
  The impressions will be scanned to provide a gold standard reference STL files.
  Interventions: Device: conventional impression stone casts digitization
- optical impressions with additional geometric scanning aids coupled with the scan bodies (Experimental): Nine optical impressions will be obtained while additional geometric scanning aids are coupled with the scan bodies to get nine CAD/CAM 3D-printed polymer casts with digital implant analogs.
  Interventions: Device: digital scanning with coupled scanning aiding device; Device: Digital Implant Model assessment of accuracy

INTERVENTIONS:
Device: conventional impression stone casts digitization — Nine conventional physical open tray impressions will be poured into a hard dental stone to obtain nine definitive implant casts with conventional implant analogs to act as a reference comparator.
  Impressions will be digitized to reference STL files.
  Arms: conventional physical impressions
Device: digital scanning with coupled scanning aiding device — Nine optical impressions will be obtained while additional geometric scanning aids are coupled with the scan bodies to get nine CAD/CAM 3D-printed polymer casts with digital implant analogs.
  Arms: optical impressions with additional geometric scanning aids coupled with the scan bodies
Device: Digital Implant Model assessment of accuracy — The nine STL files of optical scanning will serve as reference data for comparison with the digitized DIMs to evaluate the accuracy of representation of the actual position of implants in the software.
  Arms: optical impressions with additional geometric scanning aids coupled with the scan bodies

SUMMARY:
The goal of this clinical trial study is to evaluate the accuracy of the full digital workflow for four-implant, screw-retained mandibular hybrid prostheses in patients with completely edentulous mandible.

DETAILED DESCRIPTION:
The main issues to evaluate are:

* The trueness of full arch digital scans when additional geometric scanning aids are coupled with the scan bodies.
* The trueness of the generated 3D-printed DIMs.

Participants will provide two types of impressions to compare after osteointegration; the first will be conventional open tray impression used as a gold standard comparator, the second will be digital scans with additional geometric scanning aids coupled with the scan bodies.

Accordingly generated 3D-printed DIMs will be printed and compared to the digital image to evaluate its accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Patients having a completely edentulous lower arch that could be restored by fixed screw-retained implant hybrid dentures.
* Patients having a substantial bone height and width at prospective implant sites to install four standard-size inter-foraminal implants.
* Sufficient crown height space according to criteria of all-on-4.
* good oral hygiene and motivation

Exclusion Criteria:

* Patients with bad oral hygiene.
* Patients with limited mouth opening.
* Vulnerable groups.
* Uncooperative patients.
* Patients receiving or undergoing radiotherapy or chemotherapy.
* Patients with systemic diseases affecting bone metabolism.
* Smokers

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Trueness of full arch digital scans when additional geometric scanning aids are coupled with the scan bodies. | 2 months
  The optical impressions will be obtained by an intraoral scanner while the scan abutments are coupled with 3D geometric scanning aids and seated in positions.
  special digital software will be used to compare the trueness of virtual implant positions in the obtained digital scan STL files to the digitized reference positions in the patients' digitized conventional stone model

SECONDARY OUTCOMES:
Trueness of the generated 3D-printed digital implant models. | 2 months
  Based on the obtained optical scans, CAD software will be used to produce CAM files of definitive implant casts, the polymer casts will be printed and the digital implant analogs will be installed in their corresponding positions in the printed DIMs.
  The digitized data of the DIMs will be compared to their corresponding reference STL files of optical scans to check the accuracy of the generated digital implant models.